CLINICAL TRIAL: NCT03168555
Title: Changes in Bile Acid Homeostasis and Stool Habits After Cholecystectomy
Acronym: BACH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-434; 2016-004692-53 (EudraCT Number)
Record Dates: First submitted 2017-05-22; First posted 2017-05-30 (Actual); Results first posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2021-07

CONDITIONS: Bile Acid Malabsorption; Cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Chenodeoxycholic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): chenodeoxycholic acid 1250mg po.
  Interventions: Drug: chenodeoxycholic acid

INTERVENTIONS:
Drug: chenodeoxycholic acid — 1250 mg CDCA is given with a study meal
  Other Names: CDCA; chenodeoxycholate

SUMMARY:
Investigate serial plasma samples of fibroblast growth factor 19 (FGF19) after oral stimulation with chenodeoxycholic acid in the same subjects before and after elective cholecystectomy

DETAILED DESCRIPTION:
Lack of FGF19 and elevated 7-alpha-hydroxy-colestenone (C4) is associated with the bile acid diarrhoea (BAD), a disease with increasing estimated of prevalence.

BAD is occasionally triggered by cholecystectomy and FGF19 and C4 is known to be affected by cholecystectomy. The investigators are exploring if FGF19 after oral stimulation can be developed to a universal test for BAD, and need to know how the proposed test is affected by cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* planned elective cholecystectomy

Exclusion Criteria:

* small bowel resection
* right sided hemicolectomy
* known chronic diarrheal disease (celiac disease, lactose malabsorption, Inflammatory bowel diseases, incl microscopic colitis)
* pregnancy
* wish for pregnancy within next three months
* allergy to eggs
* allergy to constituents in Xenbilox (capsules with chenodeoxycholic acid)
* acute cholecystitis within two months
* chronic cholecystitis
* cirrhosis of the liver
* suspected obstructive choledocholithiasis
* icterus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-06-22 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Borup, Principal Investigator — Zealand University Hosipital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Visit 1 (Pro-operative)
Arm/Group | Intervention
Started | 23
Completed | 22
Not Completed | 1
Not completed — intercurrent disease, drop-out before visit 1 | 1
Period: Visit 2 (Post-operative)
Arm/Group | Intervention
Started | 22
Completed | 18
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 23 patients enrolled but one dropped out before visit 1. Baseline characteristics therefore only are available for 22
Arm/Group | Intervention
Number analyzed (Participants) | 22
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [38 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 22
Region of Enrollment [Number; unit: participants]
  Denmark | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Stimulated Fibroblast Growth Factor 19 (FGF19) From Baseline Before Versus Post Cholecystectomy
Description: Change from baseline to after cholecystectomy in median chenodeoxycholic acid (CDCA) plus meal stimulated FGF19 (delta 0 min to 150 min after stimulation)
Time Frame: baseline and 3 - 5 months after cholecystectomy
Measure: Median (Inter-Quartile Range); unit: pg per mL
Groups:
- Visit 1; Visit 2: chenodeoxycholic acid 1250mg po.
  chenodeoxycholic acid: 1250 mg CDCA is given with a study meal
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
pg per mL | 81 [-20 to 274] | 186 [111 to 382]
Statistical Analysis 1: Comparison: Visit 1 vs Visit 2; Test type: Equivalence — compares visit 1 with visit 2; p = 0.03, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in Chenodeoxycholic Acid (CDCA) Absorption to Plasma From Baseline Before Versus After Cholecystectomy
Description: Change from baseline to after cholecystectomy in median unconjugated CDCA plus meal stimulated absorption of unconjugated CDCA to measured in plasma (total area under the CDCA curve with measurement at fasting ie. t=0 minutes and subsequently at 60, 90, 120, and finally at 150minutes.
Time Frame: baseline and 3 - 5 months after cholecystectomy
Population: compares visit 1 with visit 2
Measure: Median (Inter-Quartile Range); unit: µM * minutes
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
µM * minutes | 1554 [1084 to 2231] | 1847 [1310 to 2193]

3. Secondary Outcome: Change in Fasting 7-alpha-hydroxy-cholestenone (C4) From Baseline Before Versus After Cholecystectomy
Description: Change from baseline to after cholecystectomy in fasting C4
Time Frame: baseline and 3 - 5 months after cholecystectomy
Population: paired t-test of lognormalized values
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
ng/mL | 6.0 [4.1 to 8.7] | 7.5 [5.5 to 10.0]
Statistical Analysis 1: Comparison: Visit 1 vs Visit 2; compares visit 1 with visit 2; Test type: Equivalence — compares visit 1 with visit 2; p = 0.63, paired t-test; lognormalized values

4. Secondary Outcome: Change in Lipid Status From Baseline Before Versus After Cholecystectomy
Description: Change from baseline to after cholecystectomy in plasma triglycerides
Time Frame: baseline and 3 - 5 months after cholecystectomy
Population: visit 1 compared with visit 2
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
mmol/L | 1.4 [1.1 to 2.1] | 1.5 [1.1 to 1.9]
Statistical Analysis 1: Comparison: Visit 1 vs Visit 2; Test type: Superiority; p = 0.32, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Change in Stool Frequency From Baseline Before Versus After Cholecystectomy
Description: Change from baseline to after cholecystectomy in number of stools as a mean of a seven-day diary baseline versus after cholecystectomy. That is the diary results for each study participant is tallied using mean values. The tallying of these diary results is done using medians. Therefore the unit used is 'mean stools per day' and this is reported with medians
Time Frame: baseline and 3 - 5 months after cholecystectomy
Measure: Median (Inter-Quartile Range); unit: mean stools per day
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
mean stools per day | 1.6 [1.1 to 2.0] | 1.6 [1.3 to 1.7]
Statistical Analysis 1: Comparison: Visit 1 vs Visit 2; Test type: Superiority; p = 0.73, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Change in Stool Pattern Correlated to FGF19
Description: Spearman correlation between change from baseline to after cholecystectomy in FGF19 and in mean number of stools
Time Frame: baseline and 3 - 5 months after cholecystectomy
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Intervention
Number analyzed (Participants) | 18
Spearman correlation coefficient | -0.21
Statistical Analysis 1: Comparison: Intervention; Test type: Other — Spearman correlation; p = 0.41, Spearman correlation

7. Secondary Outcome: Change in Patient Reported Diarrhea Symptoms Correlated With Change in C4 From Baseline Before Versus After Cholecystectomy
Description: Correlation between patient reported frequency of diarrhea (gastrointestinal quality of life index item 31) and fasting C4 before versus after cholecystectomy
Time Frame: baseline and 3 - 5 months after cholecystectomy
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
Spearman correlation coefficient | -.23 | -0.52
Statistical Analysis 1: Comparison: Visit 1; Test type: Other — Spearman correlation; p = 0.35, Spearman correlation
Statistical Analysis 2: Comparison: Visit 2; Test type: Other; p = 0.03, Spearman correlation

8. Secondary Outcome: Change in C4 Total Area Under the Curve From Baseline Before Versus After Cholecystectomy
Description: Change in total AUC for C4 between visit 1 and visit 2
Time Frame: before cholecystectomy and 3-5 months after cholecystectomy
Measure: Mean (95% Confidence Interval); unit: ng/mL x minutes
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
ng/mL x minutes | 774 [524 to 1143] | 1040 [765 to 1417]
Statistical Analysis 1: Comparison: Visit 1 vs Visit 2; Test type: Equivalence — comparing visit 1 with visit 2; p = 0.36, paired t-test

9. Secondary Outcome: Change in Fasting FGF19 From Baseline Before Versus After Cholecystectomy
Description: change in fasting FGF19 before versus after cholecystectomy
Time Frame: before and 3-5 months after cholecystectomy
Measure: Mean (95% Confidence Interval); unit: pg per mL
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
pg per mL | 102 [74 to 141] | 92 [67 to 125]
Statistical Analysis 1: Comparison: Visit 1 vs Visit 2; Test type: Superiority; p = 0.29, paired t-test

10. Secondary Outcome: Change in Patient Reported Diarrhea Symptoms Correlated With Change in FGF19 From Baseline Before Versus After Cholecystectomy
Description: Correlation between patient reported frequency of diarrhea (gastrointestinal quality of life index item 31) and fasting FGF19 before versus after cholecystectomy
Time Frame: baseline and 3 - 5 months after cholecystectomy
Measure: Number; unit: Spearman correlation coefficient
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
Spearman correlation coefficient | 0.08 | -0.07
Statistical Analysis 1: Comparison: Visit 1; Test type: Other — Spearman correlation; p = 0.73, Spearman correlation
Statistical Analysis 2: Comparison: Visit 2; Test type: Other; p = 0.77, Spearman correlation

11. Secondary Outcome: Change in Stool Consistency (Bristol Stool Type) From Baseline Before Versus After Cholecystectomy
Description: Change from baseline to after cholecystectomy in mean Bristol type per stool as of a seven-day diary baseline versus after cholecystectomy. The Bristol scale divides stool into seven categories from 1 (hard lumps) to 7 (completely watery stool). The diary shows pictograms with short text descriptions.
Time Frame: baseline and 3 - 5 months after cholecystectomy
Measure: Median (Inter-Quartile Range); unit: Bristol stool type
Arm/Group | Visit 1 | Visit 2
Number analyzed (Participants) | 18 | 18
Bristol stool type | 4.2 [3.7 to 4.8] | 4.0 [3.6 to 4.5]
Statistical Analysis 1: Comparison: Visit 1 vs Visit 2; Test type: Superiority; p = 0.80, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were registered in relation to administration of chenodeoxycholic acid both at visit 1 and visit 2 (separated by 3-5 months). Registration started at time of administration of chenodeoxycholic acid (one dose) and the registration lasted four days after this. At day three after the administration standard liver biochemistry was measured (ALT, Alk. phospatase, INR, bilirubin).
Arm/Group | Visit 1 | Visit 2
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/18
Other Adverse Events (participants affected / at risk) | 22/22 | 15/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Visit 1 (N=22) | Visit 2 (N=18)
Headache (Nervous system disorders) | 1 (1) | 0 (0) — SNOMED CT: 25064002
Migraine (Nervous system disorders) | 1 (1) | 0 (0) — SNOMED CT: 37796009
Dizzyness (Nervous system disorders) | 1 (1) | 0 (0) — SNOMED CT: 404640003
Fatigue (General disorders) | 2 (2) | 0 (0) — SNOMED CT:224960004
Abdominal bloating (Gastrointestinal disorders) | 1 (1) | 1 (1) — SNOMED CT: 116289008
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) — SNOMED CT: 422587007
Diarrhea (Gastrointestinal disorders) | 14 (14) | 14 (14) — SNOMED CT:62315008
Burping (Gastrointestinal disorders) | 1 (1) | 0 (0) — SNOMED CT: 271834000
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 5 (5) — SNOMED CT: 21522001
Heartburn (Gastrointestinal disorders) | 1 (1) | 1 (1) — SNOMED CT:16331000
Malaise (General disorders) | 1 (1) | 0 (0) — SNOMED CT:367391008
Abdominal sounds/growling (Gastrointestinal disorders) | 5 (5) | 2 (2) — SNOMED CT: 249503000

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/55/NCT03168555/Prot_SAP_000.pdf